CLINICAL TRIAL: NCT06595147
Title: Breast cancEr, FITness and ExeRcise for Heart Health: The BE-FITTER Study
Acronym: BE-FITTER
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Alberta (Other)
Collaborators: Canadian Institutes of Health Research (CIHR) (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: HREBA.CC-24-0058
Record Dates: First submitted 2024-05-06; First posted 2024-09-19 (Actual); Last update posted 2026-01-08 (Actual); Status verified 2026-01

CONDITIONS: Breast Cancer; Disability Physical; Heart Failure; Cardiotoxicity
Keywords: Exercise Training; Fitness; Heart; Muscle; Cancer; Survivorship
MeSH Terms: conditions — Breast Neoplasms; Heart Failure; Cardiotoxicity; Neoplasms

STUDY DESIGN:
Who Masked: Outcomes Assessor
Masking Description: All MRI outcomes will be performed blinded to group allocation. Outcome assessors for post-outcome assessments will be blinded to baseline values.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental Arm: Structured Exercise Training (Experimental): Participants randomized to exercise training will be provided with a 12-week structured exercise training program. The program includes 3 weekly sessions of aerobic exercise (e.g treadmill, cycling, elliptical machine) and/or resistance training (i.e lifting weights). The aerobic sessions will include long-endurance (40-60 minutes at moderate intensity), tempo (30-40 minutes at a moderate-vigorous intensity) and high-intensity interval exercise (10-15 intervals of 30-60 seconds at 100% peak aerobic power output, interspersed with 60 seconds of active recovery). Resistance training will include 4-6 lower body exercises performed for 2-3 sets of 8-20 repetitions at a load equivalent to 60-85% of their one repetition maximum. The program will be supervised by an exercise trainer (Clinical Exercise Physiologist, Physiotherapist, Kinesiologist or Research Associate with exercise training experience) and will be individualized each individual's baseline fitness and medical history.
  Interventions: Behavioral: Structured Exercise Training
- Active Comparator: Group-based Yoga and Stretching (Active Comparator): Participants allocated to the yoga and stretching group will provided with a once weekly yoga and stretching group class. The classes will consist of a combination of light-intensity yoga, balance and stretching exercises. The yoga and stretching class will be overseen by a yoga instructor, physiotherapist, physiotherapy trainee or research assistant with exercise training background
  Interventions: Behavioral: Group-based Yoga and Stretching

INTERVENTIONS:
Behavioral: Structured Exercise Training — Participants will complete 12-weeks of supervised, structured moderate-to-high intensity aerobic and resistance training three times per week.
  Arms: Experimental Arm: Structured Exercise Training
Behavioral: Group-based Yoga and Stretching — Participants will complete 12-weeks of supervised group-based yoga and stretching once per week.
  Arms: Active Comparator: Group-based Yoga and Stretching

SUMMARY:
The chemotherapy medications used for breast cancer treatment are important for achieving a cure, but a potential side effect is that they can cause a decline in functional capacity (reduced exercise tolerance and impaired physical function) and increase the risk of cardiovascular disease. The risks of decreased functional capacity and cardiovascular disease are highest in breast cancer survivors as they grow older. The factors causing the decline in functional capacity are not well understood, however they may be related to a reduction in cardiac function (e.g. decreased pumping ability of the heart) or skeletal muscle function (reduced muscle blood flow and oxygenation). Exercise training is used for other populations at risk for cardiovascular disease (such as cardiac rehabilitation), but is not routinely offered to breast cancer survivors. Therefore this research study wants to test whether exercise training can improve heart and muscle health, and increase functional capacity in up to 60 older breast cancer survivors aged >60 years old who previously received chemotherapy drugs that can affect the heart.

The purpose of this study is to compare two rehabilitation approaches: a 12-week structured exercise training program or a 12-week stretching-yoga program. The investigators want to compare whether these programs can improve functional capacity, and heart and skeletal muscle function. To do this, some of the participants in this study will be randomly enrolled in the structured exercise training program and others will be randomly enrolled in the stretching-yoga program.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥60 years
* Previously diagnosed with early-stage (I-III) BC
* Completed (≥1 year post) primary cardiotoxic treatment (anthracycline-based chemotherapy or trastuzumab-based biological therapy).

Exclusion Criteria:

* Have a history of coronary artery disease, heart failure, persistent and permanent arrhythmia (e.g. currently in atrial fibrillation), stroke, or chronic obstructive pulmonary disease
* Develop signs or symptoms of myocardial ischemia (≥1mm horizontal or down-sloping ST segment depression on electrocardiogram) during the cardiopulmonary (VO2peak) test
* Have any research MRI contraindications (e.g. any type of pacemaker), or any orthopedic limitation preventing exercise testing
* Currently performing structured exercise training (defined as ≥30 mins/day of moderate-to-vigorous aerobic and/or resistance exercise training on ≥4 days/week)
* Are unwilling to be randomized to either ExT or STRETCH

Min Age: 60 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2024-07-01 (Actual); Primary Completion 2026-12-20 (Estimated); Study Completion 2026-12-20 (Estimated)

PRIMARY OUTCOMES:
Peak arterio-venous oxygen content difference | 12 Weeks
  Peak exercise arterio-venous oxygen content difference assessed using whole-body exercise MRI
Peak cardiac output | 12 Weeks
  Peak exercise cardiac output assessed using whole-body exercise MRI

SECONDARY OUTCOMES:
Peak volume of oxygen uptake | 12 Weeks
  Peak volume of oxygen uptake assessed from a maximal cardiopulmonary exercise test
Peak diffusive muscle oxygen conductance | 12 Weeks
  Calculated diffusive muscle oxygen conductance assessed using whole-body exercise MRI
Peak stroke volume | 12 Weeks
  Peak exercise stroke volume assessed using whole-body exercise MRI
Aerobic endurance | 12 Weeks
  Walk distance measured during a six minute walk test
Physical Function | 12 Weeks
  Short physical performance battery total score (Score from 0 to 12, where higher scores represent better function)
Skeletal muscle volume | 12 Weeks
  Muscle volume of the thigh and lower leg from MRI
Skeletal muscle myosteatosis | 12 Weeks
  Muscular fat fraction of the thigh and lower leg from MRI
Skeletal muscle fibrosis | 12 Weeks
  Muscular fibrosis of the thigh and lower leg measured from MRI T1 values
Calf muscle aerobic capacity | 12 Weeks
  Peak muscle oxygen uptake from maximal plantar flexion exercise MRI
Calf muscle oxygen extraction | 12 Weeks
  Peak muscle arterio-venous oxygen difference from maximal plantar flexion exercise MRI
Calf muscle oxygen diffusive conductance | 12 Weeks
  Peak muscle oxygen diffusive conductance from maximal plantar flexion exercise MRI
Calf muscle metabolism | 12 Weeks
  Exercise phosphate and phosphocreatine responses during plantar flexion exercise 31P magnetic resonance spectroscopy
10-year Framingham Risk Score | 12 Weeks
  10-year Framingham Risk Score will be calculated from participant Sex, Age, HDL-cholesterol, Total Cholesterol, Resting Systolic Blood Pressure, Smoking Status and presence of Diabetes. The score ranges from 0% to 100% where higher scores indicate higher CVD risk.

OTHER OUTCOMES:
Habitual Physical Activity | 12 Weeks
  Time spent in moderate-to-vigorous physical activity over 7 days of objective monitoring (Fitbit)
Fasting Lipids | 12 Weeks
  A fasting blood test will be used to measure concentrations of high-density lipoprotein (HDL) cholesterol, low-density lipoprotein (LDL) cholesterol, total cholesterol and triglycerides
Fasting Glycaemic Control | 12 Weeks
  A fasting blood test will be used to measure concentrations of fasting plasma glucose and fasting insulin
Fasting Insulin Resistance | 12 Weeks
  Fasting insulin resistance will be calculated from fasting plasma glucose and insulin concentrations using the Homeostatic Model Assessment of Insulin Resistance (HOMA-IR) method.
C-reactive protein | 12 Weeks
  Plasma concentrations of C-reactive protein will be assessed from a fasting blood test.
Resting blood pressure | 12 Weeks
  Resting systolic and diastolic blood pressure will be measured in the supine position using an automated oscillometric blood pressure cuff.
Functional Assessment of Cancer Therapy - Breast (FACT-B) Questionnaire | 12 Weeks
  Quality of Life, including physical, emotional and social wellbeing and breast cancer related symptom score on the FACT-B questionnaire. Participants will be scored from 0 to 148, where 148 represents the highest quality of life.

CONTACTS AND LOCATIONS:
Locations (1):
- University of Alberta, Edmonton, Alberta, Canada

IPD SHARING:
Plan to Share IPD: No